CLINICAL TRIAL: NCT03054441
Title: Detection of Asymmetries in Upper Limb Use Through Actigraphs
Brief Title: Actigraphs for Detection of Asymmetries
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other); The University of Queensland (Other); Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: GR-2011-02350053
Record Dates: First submitted 2017-02-11; First posted 2017-02-15 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Hemiplegia; Hemiplegic Cerebral Palsy
Keywords: Upper limb; Inertial sensors
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Children, Adolescents and Young with hemiplegia
  Interventions: Other: Actigraph
- Control group: Children, Adolescents and Young with typical development
  Interventions: Other: Actigraph

INTERVENTIONS:
Other: Actigraph — Actigraphs worn on wrists

SUMMARY:
In hemiplegia quantitatively measurement of the asymmetry in the use of upper limbs could overcome the limitation of many outcome measures in which scores are dependent on the experience and training of the therapist. The main aim of this study was to determine the validity of Actigraph GXT3+ to measure asymmetry in the use of the two upper limbs during the Assisting Hand Assessment (AHA) in children, adolescents and young with hemiplegia aged 5-19 years, compared to age-matched typically developing subjects (TD).

DETAILED DESCRIPTION:
This study aims to validate the use of Actigraphs as an evaluation tool of the upper limb asymmetry in children / adolescents and young adults with typical development or hemiplegia.

The validation involves two stages:

The first stage, carried out in the clinical setting, provides the use of Actigraphs (Actigraph GXT3+ and in a subgroup also FitBit) during the administration of clinical tests which are usually performed for the evaluation of the manual dominance in individuals with hemiplegia but also suitable for those with typical development.

This first phase will allow to compare the quantitative measures acquired by the actigraphs (e.g. the mean activity of each hand and the asymmetry index i.e. difference between the mean activities of the two arms) with those from clinical standardized measures.

The second phase, carried out in a non-clinical setting, provides the use of Actigraphs (Actigraph GXT3+ and in a subgroup also FitBit) in a subgroup of subject involved in the first phase for a week in order to measure the asymmetry index during the activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3-25 years
* Hemiplegia (experimental group) or Voluntary adhesion (control group)

Exclusion Criteria:

* movement disorders
* sensory deficits

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children, Adolescents and Adults with hemiplegia and age-matched controls with typical development
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Correlation between Asymmetry Index (AI) and Assisting Hand Assessment (AHA) scores. | Baseline
  The asymmetry index (AI) is the difference between the mean activities of the dominant with those of the non dominant hand and it will be correlated with the scores of AHA. The AHA measures Upper Limb function during bimanual activities. The test evaluates spontaneous use of assisting hand during a semi-structured 10-15 minutes session with specific toys (Kids-AHA) or tasks (Ad-AHA) requiring bimanual handling.

SECONDARY OUTCOMES:
Correlation between AI during AHA and AI in 7 days | Baseline- 1 week
  Correlation of AI between a standardized bimanual test with 7 days of common daily life

OTHER OUTCOMES:
Correlation between Box and Block test (BBT) and mean activity of dominant and non dominant hand | Baseline
  The mean activity of each hand will be correlated with the BBT that measures unilateral gross manual dexterity. It is a quick (2-5 minutes), simple and inexpensive test. It can be used with a wide range of populations from childhood to adulthood.
Correlation among Mean activity and asymmetry index during standardized clinical activities. | Baseline
  The mean activity of each hand and the asymmetry index will be analyzed during some other activities such as Writing, Upper Limb Physician's Rating Scale, Six Minutes Walking Test, Rest Supine Position

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Sgandurra, MD, PhD, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- IRCCS Stella Maris Foundation, Calambrone, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JL, Hakim AD. Wrist actigraphy. Chest. 2011 Jun;139(6):1514-1527. doi: 10.1378/chest.10-1872. PMID 21652563
- [Background] Nagels G, Marion P, Pickut BA, Timmermans L, De Deyn PP. Actigraphic evaluation of handedness. Electroencephalogr Clin Neurophysiol. 1996 Jun;101(3):226-32. doi: 10.1016/0924-980x(96)95566-6. PMID 8647035
- [Derived] Beani E, de 'Cavalieri MF, Filogna S, Barzacchi V, Cianchetti M, Maselli M, Martini G, Menici V, Prencipe G, Sicola E, Cioni G, Sgandurra G. Wearable sensors for measuring spontaneous upper limb use in children with unilateral cerebral palsy and typical development. J Neuroeng Rehabil. 2025 Apr 3;22(1):71. doi: 10.1186/s12984-025-01601-3. PMID 40181251
- [Derived] Beani E, Maselli M, Sicola E, Perazza S, Cecchi F, Dario P, Braito I, Boyd R, Cioni G, Sgandurra G. Actigraph assessment for measuring upper limb activity in unilateral cerebral palsy. J Neuroeng Rehabil. 2019 Feb 22;16(1):30. doi: 10.1186/s12984-019-0499-7. PMID 30795810